CLINICAL TRIAL: NCT00947973
Title: Multisite Study of School Based Treatment Approaches for ADHD Adolescents
Brief Title: Comparing School Based Interventions for Adolescents With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH082865 (NIH); R01MH067949 (NIH); 1R01MH082865-01A2 (NIH); 1R01MH082864-01A2 (NIH); DSIR 84-CTS
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; School Based; Intervention; Psychosocial; Academic Intervention; Behavioral
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Behavior | interventions — somatostatin, cyclic hexapeptide(Phe-Phe-Trp-Lys-Thr-Phe)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Challenging Horizons Program after-school model (Experimental): Participants will receive the CHP after-school model.
  Interventions: Behavioral: Challenging Horizons Program (CHP) after-school model
- Challenging Horizons Program consultation model (Experimental): Participants will receive the CHP consultation model.
  Interventions: Behavioral: Challenging Horizons Program (CHP) consultation model
- Community care (No Intervention): Participants will have access to standard community care.

INTERVENTIONS:
Behavioral: Challenging Horizons Program (CHP) after-school model — Interventions delivered by a counselor 2 days a week as an after-school program. Interventions will strengthen skills in materials organization, homework management, studying, note taking, and socialization.
  Arms: Challenging Horizons Program after-school model
Behavioral: Challenging Horizons Program (CHP) consultation model — Interventions delivered by a mentor (e.g., a teacher or school counselor) as needed, with expert consultation available
  Arms: Challenging Horizons Program consultation model

SUMMARY:
This study will compare the efficacy and cost effectiveness of two methods of treating adolescents with attention deficit hyperactivity disorder in school.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is characterized by inattention, hyperactivity, and impulsivity. Approximately 50% to 70% of children who had ADHD continue to meet its criteria in adolescence, but the problems stemming from adolescent ADHD can be more serious-including an increased risk of substance use, delinquency, academic failure, serious social impairment, and legal problems. Problems in school more than double when students with ADHD move from elementary school to middle and high school.

Treating ADHD with medications alone is often ineffective, but adding other methods, such as behavioral treatments, may be beneficial. Researchers have developed a psychosocial treatment for adolescents with ADHD, called the Challenging Horizons Program (CHP), that is delivered in school and targets social impairment, family conflict, and academic failure. Two versions of CHP were developed, an after-school model and a consultation model. The after-school model involves 2 to 3 days of individualized treatment per week and has a higher cost than the consultation model because it involves hiring specialized counseling staff and finding space to house the program after school. The consultation model involves teaching CHP intervention strategies to school staff, who then mentor students with ADHD and deliver interventions as needed to solve problems. This model is less expensive, but it does not deliver treatment as often or consistently as the after-school model. This study will compare the after-school and consultation models of the CHP to determine their relative efficacy and cost effectiveness. The study will also evaluate factors that may predict which adolescents would benefit most from either of the two models.

Participation in this study will last a full school year. Participants from schools taking part will be randomly assigned to one of three groups: after-school CHP, consultation CHP, or standard community care. Participants receiving after-school CHP will attend two 2.5-hour after-school sessions per week in which they will work with counselors on homework management, educational skills, and interpersonal skills. Participants receiving consultation CHP will be assigned a teacher mentor (who will volunteer to work with the student), and the mentor and student will meet as needed. A study clinician will provide support to the teacher mentors, who will learn the same interventions as counselors in the after-school condition. Participants in the community care condition will not receive any intervention but will receive a list of community psychosocial and medical service providers for children and their families. All participants will undergo study assessments pre-treatment; in November, January, and March of the school year; post-treatment; and at a 6-month follow-up. Assessments will include questionnaires and clinical interviews completed by student, their parents, and their teachers. ADHD symptoms, academic performance, relevant skills of adolescents, and program costs will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for ADHD, including all ADHD subtypes (predominately inattentive, predominately hyperactive/impulsive, and combined)
* All common comorbid conditions not listed as exclusionary will be included.

Exclusion Criteria:

* Full Scale Intelligence Quotient (FSIQ) less than 80
* Anticipated attendance for participant or parent less than 80% for scheduled activities
* Meets diagnostic criteria for bipolar disorder, psychotic disorder, substance dependence (but not substance abuse), or obsessive-compulsive disorder (OCD)

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 315 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Teacher ratings of academic performance on the Impairment Rating Scale | Measured pre-intervention, 3 times during the intervention, post-intervention, and at a 6-month follow-up

SECONDARY OUTCOMES:
Grade point average (GPA) | Measured pre-intervention, post-intervention, and at a 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M. Langberg, PhD, Principal Investigator — University of Cincinnati College of Medicine, Cincinnati Children's Hospital Medical Center; Steven W. Evans, PhD, Principal Investigator — Ohio University
Locations (2):
- United States (2):
  - Ohio University, Athens, Ohio
  - Cincinnati Children's Hospital Medical Center, Center for ADHD, Cincinnati, Ohio